CLINICAL TRIAL: NCT00697775
Title: Study to Assess the Feasibility of GSK Bio's Candidate HBV / MPL Vaccines Following Different Schedules and Formulations and to Compare Their Safety and Immunogenicity to That of Engerix™-B in Healthy Adolescents Aged 11 to 15
Brief Title: Safety and Immunogenicity of GSK Bio's Candidate HBV-MPL Vaccines Compared to Engerix™-B, in Healthy Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Isabelle Harpigny, GSK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 208129/028
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Last update posted 2008-06-16 (Estimated); Status verified 2008-06

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Recombinant hepatitis B vaccine; Adjuvant
MeSH Terms: conditions — Hepatitis B

ARMS (4):
- Group A (Experimental): HBV-MPL Formulation A at months 0 and 6
  Interventions: Biological: HBV-MPL vaccine Formulation A
- Group B (Experimental): HBV-MPL Formulation B at months 0 and 6
  Interventions: Biological: HBV-MPL vaccine Formulation B
- Group C (Experimental): HBV-MPL Formulation A at month 0 and Engerix™-B at month 6
  Interventions: Biological: HBV-MPL vaccine Formulation A; Biological: Engerix™-B
- Group D (Active Comparator): Engerix™-B at months 0, 1, 6
  Interventions: Biological: Engerix™-B

INTERVENTIONS:
Biological: HBV-MPL vaccine Formulation A — Single dose (when extemporaneously co-administered with Engerix™-B) or 2-dose (when administered alone) intramuscular injection
  Arms: Group A; Group C
Biological: HBV-MPL vaccine Formulation B — 2-dose intramuscular injection
  Arms: Group B
Biological: Engerix™-B — Single dose (when extemporaneously co-administered with HBV-MPL) or 3-dose (when administered alone) intramuscular injection
  Arms: Group C; Group D

SUMMARY:
In this study the safety and immunogenicity of 2 different formulations of the candidate HBV-MPL vaccine administered according to a 0, 6-month schedule were explored and compared to that of Engerix™-B in healthy adolescents aged 11 to 15

DETAILED DESCRIPTION:
At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham

ELIGIBILITY:
Inclusion Criteria:

* Age: between 11 and 15 years at the time of the first vaccination.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Written informed consent obtained from the parents or guardians of the subject and from the subject himself/herself in all subjects 15 years of age.
* If the subject is female, she must be of non-childbearing potential, if of childbearing potential, she must be abstinent or have used an adequate contraceptive for one month prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) during the study period or within 30 days preceding the first dose of study vaccine.
* Administration of chronic (defined as more than 14 days) immunosuppressants or other immune-modifying drugs within six months of vaccination.
* Planned administration of a vaccine not foreseen by the study protocol during the period starting from one week before each dose of vaccine and ending 30 days after.
* Previous vaccination against hepatitis B virus.
* Previous vaccination with vaccine containing MPL.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrollment.
* Hepatomegaly, right upper quadrant abdominal pain or tenderness.
* Axillary temperature of ≥ 37.5° C.
* Administration of immunoglobulin and / or any blood product within the six months preceding the first dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* History of chronic disease deemed by the investigator to be relevant.
* Positive for anti-HBV antibodies at screening

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 1998-03; Primary Completion 1999-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of Serious adverse experiences (SAE) | During the study period
Occurrence, intensity and relationship to vaccination of solicited local and general symptoms | During the 8-day follow-up period after vaccination
Occurrence, intensity and causal relationship of unsolicited adverse events | 31-day follow-up period after vaccination

SECONDARY OUTCOMES:
Anti-HBs antibody concentrations | At months 1, 2, 6, and 7
Cell mediated immunity | At months 1, 6, and 7

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Clinical Trials Call Center, Mainz, Germany